CLINICAL TRIAL: NCT03592771
Title: Communication App to Manage Symptoms and Improve Adjuvant Endocrine Therapy Adherence
Brief Title: THRIVE Breast Cancer App Study
Acronym: THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); West Cancer Center (Other); Vector Oncology (Other)
Responsible Party: Principal Investigator, Ilana Graetz, Associate Professor, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00109957; 1R01CA218155 (NIH)
Record Dates: First submitted 2018-07-05; First posted 2018-07-19 (Actual); Results first posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Breast Neoplasm Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Participants use an electronic pill monitoring device with their AET medication and complete a survey at baseline and again after 12 months.
- THRIVE App (Active Comparator): Participants use a web-based app to report their AET use in the previous 7 days and any treatment-related symptoms or changes in the severity of symptoms. Participants receive reminders via text or email to use the app once per week during the 6-month intervention phase. Participants use an electronic pill monitoring device with their AET medication and complete a survey at baseline and again after 12 months.
  Interventions: Behavioral: THRIVE App
- THRIVE App+Feedback (Active Comparator): Participants use a web-based app to report their AET use in the previous 7 days and any treatment-related symptoms or changes in the severity of symptoms. Participants receive reminders via text or email to use the app once per week during the 6-month intervention phase. In addition, participants in this group will also receive weekly tailored feedback text messages or images during the 6-month intervention phase. Participants use an electronic pill monitoring device with their AET medication and complete a survey at baseline and again after 12 months.
  Interventions: Behavioral: THRIVE App; Behavioral: Tailored Feedback Messages

INTERVENTIONS:
Behavioral: THRIVE App — Participants in the THRIVE App group receive a weekly text message to prompt them to log into the THRIVE app to answer questions about their AET adherence and related adverse symptoms. The app can be accessed through any web-enabled device or Internet browser. All participant-reported data will be automatically entered into the patient's electronic health record and easily available to the care team for review. Any concerning symptoms or changes will trigger an email alert to the patient's oncology team.
  Arms: THRIVE App; THRIVE App+Feedback
Behavioral: Tailored Feedback Messages — Participants receive weekly tailored feedback messages and/or images based on their baseline survey responses and use of the app during the 6-month intervention phase. Some tailored feedback includes links to symptom-specific educational materials and coping strategies for participants who report low-severity symptoms. Message categories are tailored to participant's responses to the app and baseline survey.
  Arms: THRIVE App+Feedback

SUMMARY:
This study will test the use of a web-enabled app that is integrated directly with patients' electronic health records, with and without tailored feedback. The app-based intervention is designed to improve patient-provider communication outside of clinic visits, resulting in improved symptom management and adjuvant endocrine therapy adherence among diverse patients with hormone receptor-positive breast cancer. The researchers will evaluate the impact of the intervention on a comprehensive set of outcomes, including rigorous measures of long-term adherence, quality of life, and costs.

DETAILED DESCRIPTION:
For women with hormone receptor-positive breast cancer, long-term use of adjuvant endocrine therapy (AET) significantly reduces the risk of hospitalizations, cancer recurrence and mortality, and increases quality of life. Despite the known benefits of AETs, many patients are nonadherent due to adverse side effects. Furthermore, lower AET adherence among black women may be contributing to the large and growing disparities in mortality outcomes. Real-time monitoring of treatment-related adverse symptoms and adherence could result in more effective management of symptoms, higher medication adherence, and ultimately lower recurrence and mortality. To date, however, only a few interventions have aimed to improve AET adherence, even fewer have targeted symptom management as a means to improve adherence, and none have found a statistically significant improvement on adherence. This study will fill this research gap by testing a web-enabled app designed with the explicit goal of improving long-term AET adherence. Patient-reported symptoms will be integrated directly with the patient's electronic health record, and concerning reports will trigger an alert to the patient's care team in order to improve timely patient-provider communication and care outside of clinic visits. In a small pilot trial of the study app, the researchers found that participants who had recently initiated a new AET and received weekly reminders to use the app reported significantly higher adherence to AETs at 8 weeks compared with a control group (91% vs. 68%, p=0.02). The proposed study builds on the success of the pilot by: 1) expanding the intervention period to six months in order to capture later-onset adverse symptoms that are slower to develop; 2) following participants for one to three years, depending on enrollment year, to test longer-term effects of the intervention on medication adherence and other outcomes; 3) including a larger sample powered to test multiple levels of the intervention; and 4) race-stratifying to test for a differential impact by race. This study will randomize 360 participants to one of three arms: 1) an "App" group (n=120) that will receive weekly reminders to use the study app; 2) an "App+Feedback" group (n=120) that will receive weekly reminders and personalized feedback based on their use of the app; or 3) a "Usual Care" group (n=120) that will receive usual care only. The app will include questions about AET adherence and adverse symptoms with built-in alerts sent to the patient's care team if any concerning symptoms or trends are reported. The researchers hypothesize that monitoring symptoms and adherence with actionable alerts and tailored feedback reports to patients will result in timelier symptom management and higher long-term adherence to AET. By evaluating the impact of the intervention on a comprehensive set of measures, including AET adherence, patient outcomes, racial disparities and resource use-related costs, this study will provide valuable and actionable results for providers, policy makers, and insurers who strive to achieve the "Triple Aim" - reduce costs while improving health outcomes and the patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients (age≥18)
* Diagnosis of ductal carcinoma in situ or Stage I-III hormone receptor-positive breast cancer
* New prescription for an aromatase inhibitor or tamoxifen
* Have a mobile device with a data plan or a home computer with Internet
* Have a valid email address
* Willing to complete brief surveys on a web-enabled device
* AET is indicated as standard of care

Exclusion Criteria:

* Unable to communicate in English
* Prior use of adjuvant endocrine therapy (aromatase inhibitor or tamoxifen) for current diagnosis
* Concurrently undergoing surgery, chemotherapy or radiation
* Current diagnosis of rheumatoid arthritis
* Chronic daily narcotic usage
* Patient plans to move or transfer their care within the next year

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Graetz, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - West Cancer Center, Midtown, Memphis, Tennessee
  - West Cancer Center, East Memphis, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paladino AJ, Anderson JN, Krukowski RA, Waters T, Kocak M, Graff C, Blue R, Jones TN, Buzaglo J, Vidal G, Schwartzberg L, Graetz I. THRIVE study protocol: a randomized controlled trial evaluating a web-based app and tailored messages to improve adherence to adjuvant endocrine therapy among women with breast cancer. BMC Health Serv Res. 2019 Dec 19;19(1):977. doi: 10.1186/s12913-019-4588-x. PMID 31856812
- [Derived] Graetz I, Hu X, Krukowski RA, Anderson JN, Stepanski E, Vidal G, Waters TM, Schwartzberg LS. Adherence to oral endocrine therapy by menopausal status: post hoc insights from a remote monitoring randomized trial. NPJ Breast Cancer. 2026 Jan 28. doi: 10.1038/s41523-026-00900-9. Online ahead of print. PMID 41605963
- [Derived] Hu X, Krukowski RA, Stepanski E, Anderson JN, Vidal GA, Torres MA, Schwartzberg LS, Graetz I. Racial Differences in Symptom Burden and Endocrine Therapy Adherence in Breast Cancer: A Post Hoc Analysis of a Randomized Trial. J Natl Compr Canc Netw. 2025 Sep 26;23(10):e257054. doi: 10.6004/jnccn.2025.7054. PMID 41005350
- [Derived] Graetz I, Hernandez S, Hu X, Krukowski RA, Anderson JN, Waters TM, Stepanski E, Vidal GA, Schwartzberg LS. Addressing health literacy gaps in adjuvant endocrine therapy adherence: Post hoc insights from a randomized remote monitoring trial. Breast. 2025 Oct;83:104552. doi: 10.1016/j.breast.2025.104552. Epub 2025 Aug 5. PMID 40779883
- [Derived] Arshad S, Hu X, Krukowski RA, Waters TM, Vidal GA, Schwartzberg L, Lipscomb J, Graetz I. COVID-19-Related Financial Hardship and Adherence to Adjuvant Endocrine Therapy Among Women With Early-Stage Breast Cancer. Health Serv Res. 2025 Jun 17:e14658. doi: 10.1111/1475-6773.14658. Online ahead of print. PMID 40525537
- [Derived] Krukowski RA, Hu X, Arshad S, Anderson JN, Stepanski E, Vidal GA, Schwartzberg LS, Graetz I. Symptom Monitoring App Use Associated With Medication Adherence Among Woman Survivors of Breast Cancer on Adjuvant Endocrine Therapy. JCO Clin Cancer Inform. 2024 Dec;8:e2400179. doi: 10.1200/CCI-24-00179. Epub 2024 Dec 6. PMID 39642329
- [Derived] Graetz I, Hu X, Kocak M, Krukowski RA, Anderson JN, Waters TM, Curry AN, Robles A, Paladino A, Stepanski E, Vidal GA, Schwartzberg LS. Remote Monitoring App for Endocrine Therapy Adherence Among Patients With Early-Stage Breast Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2417873. doi: 10.1001/jamanetworkopen.2024.17873. PMID 38935379

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from West Cancer Centers in East Memphis and Midtown, Memphis, Tennessee, USA. Participant enrollment began November 15, 2018 and all follow-up assessments were completed by June 30, 2022.
Groups:
- Usual Care: Participants with early-stage, hormone receptor positive breast cancer used an electronic pill monitoring device with their adjuvant endocrine therapy (AET) medication and completed a survey at baseline and again after 12 months.
- THRIVE App: Participants with early-stage, hormone receptor positive breast cancer used a web-based app to report their AET use in the previous 7 days and any treatment-related symptoms or changes in the severity of symptoms. Participants received reminders via text or email to use the app once per week during the 6-month intervention phase. Participants used an electronic pill monitoring device with their AET medication and completed a survey at baseline and again after 12 months.
- THRIVE App+Feedback: Participants with early-stage, hormone receptor positive breast cancer used a web-based app to report their AET use in the previous 7 days and any treatment-related symptoms or changes in the severity of symptoms. Participants received reminders via text or email to use the app once per week during the 6-month intervention phase. In addition, participants in this group also received weekly tailored feedback text messages or images during the 6-month intervention phase. Participants used an electronic pill monitoring device with their AET medication and completed a survey at baseline and again after 12 months.
Period: Overall Study
Arm/Group | Usual Care | THRIVE App | THRIVE App+Feedback
Started | 104 | 98 | 102
Completed | 97 | 84 | 85
Not Completed | 7 | 14 | 17
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Death | 0 | 1 | 1
Not completed — Lost to Follow-up | 5 | 11 | 15
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | THRIVE App | THRIVE App+Feedback | Total
Number analyzed (Participants) | 104 | 98 | 102 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (11.4) | 59.4 (10.3) | 58.1 (10.7) | 58.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 98 | 102 | 304
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 3 | 9
  Not Hispanic or Latino | 100 | 95 | 98 | 293
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 2 | 2 | 5
  Black or African American | 37 | 33 | 32 | 102
  White | 65 | 61 | 68 | 194
  Other | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 104 | 98 | 102 | 304
Income [Count of Participants; unit: Participants]
  <100% Federal Poverty Level (FPL) | 12 | 13 | 7 | 32
  100 to 200% FPL | 12 | 9 | 12 | 33
  201 to 400% FPL | 23 | 20 | 23 | 66
  >400% FPL | 52 | 54 | 56 | 162
  Missing | 5 | 2 | 4 | 11
Education [Count of Participants; unit: Participants]
  High school or less | 19 | 18 | 23 | 60
  More than high school | 85 | 80 | 79 | 244
Marital Status [Count of Participants; unit: Participants]
  Married or living with partner | 72 | 62 | 68 | 202
  Other | 32 | 36 | 34 | 102

OUTCOME MEASURES:

1. Primary Outcome: Adjuvant Endocrine Therapy (AET) Medication Adherence
Description: Medication adherence with prescribed AET (aromatase inhibitor or tamoxifen) is captured using an electronic monitoring pillbox (Wisepill).
Time Frame: Up to Month 12
Population: This analysis includes participants who completed the 12 month follow-up assessment.
Measure: Mean (Standard Deviation); unit: percentage of prescribed doses taken
Arm/Group | Usual Care | THRIVE App | THRIVE App+Feedback
Number analyzed (Participants) | 97 | 84 | 85
percentage of prescribed doses taken | 77 (26) | 73 (28) | 71 (30)

2. Secondary Outcome: 19 Item Endocrine Symptom Subscale (ESS-19) Score of the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES)
Description: Relative changes in adverse symptom burden were assessed using the Endocrine Symptom Subscale of the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) questionnaire. The FACT-ES is a 46-item questionnaire asking participants to report how much they have been impacted by a variety of symptoms on a 5-point scale where 0 = not at all and 4 = very much. The Endocrine Symptom Subscale consists of 19 items with total raw scores ranging from 0 to 76. Higher scores indicate greater impact from symptoms.
Time Frame: Baseline, Month 12
Population: This analysis includes participants completing the indicated study visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | THRIVE App | THRIVE App+Feedback
Number analyzed (Participants) | 104 | 98 | 102
score on a scale
  Baseline | 62.95 (9.89) | 63.01 (9.62) | 63.47 (9.23)
  Month 12: number analyzed (Participants) | 97 | 84 | 85
  Month 12 | 60.14 (11.82) | 59.29 (11.49) | 60.54 (11.26)

3. Secondary Outcome: Short Form Health Survey (SF-12) Physical Component Summary (PCS) Score
Description: Quality of life was measured with the SF-12 instrument. The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. SF-12 is a standardized self-report questionnaire that assesses mental and physical functioning. The SF-12 consists of 12 items with a Likert-type response format that measures quality of life with a Physical Component Summary (PCS) and Mental Component Summary (MCS). Subscales associated with the PCS include physical functioning, role limitations due to physical problems, bodily pain, and general health perceptions. A scoring algorithm is used to generate a total score for the PCS component that ranges from 0 to 100. Low values represent a poor health state while high values represent a good health state.
Time Frame: Baseline, Month 12
Population: This analysis includes participants who completed the indicated study visit and had no missing responses in this survey. Some participants were administered the survey but skipped questions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | THRIVE App | THRIVE App+Feedback
Number analyzed (Participants) | 103 | 97 | 101
score on a scale
  Baseline | 44.30 (10.14) | 44.87 (9.79) | 43.99 (9.65)
  Month 12: number analyzed (Participants) | 95 | 79 | 81
  Month 12 | 44.69 (10.83) | 47.57 (10.02) | 45.25 (10.32)

4. Secondary Outcome: Short Form Health Survey (SF-12) Mental Component Summary (MCS) Score
Description: Quality of life was measured with the SF-12 instrument. The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. SF-12 is a standardized self-report questionnaire that assesses mental and physical functioning. The SF-12 consists of 12 items with a Likert-type response format that measures quality of life with a Physical Component Summary (PCS) and Mental Component Summary (MCS). Subscales associated with the MCS include vitality (energy and fatigue), social functioning, role limitations due to emotional problems, and mental health. A scoring algorithm is used to generate a total score for the MCS component that ranges from 0 to 100. Low values represent a poor health state while high values represent a good health state.
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | THRIVE App | THRIVE App+Feedback
Number analyzed (Participants) | 103 | 97 | 101
score on a scale
  Baseline | 50.66 (9.59) | 50.76 (9.86) | 50.68 (10.02)
  Month 12: number analyzed (Participants) | 95 | 79 | 81
  Month 12 | 51.77 (8.38) | 49.98 (10.48) | 51.95 (9.64)

5. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Symptoms Score
Description: Relative changes in adverse symptom burden were measured using the 4-item PROMIS Self-Efficacy for Managing Symptoms short form questionnaire. Participants indicate how confident they are that they can manage their symptoms on a 5-point scale where 1 = not confident at all and 5 = very confident. Total scores range from 4 to 20 and higher scores indicate greater self-efficacy for managing symptoms.
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | THRIVE App | THRIVE App+Feedback
Number analyzed (Participants) | 102 | 98 | 102
score on a scale
  Baseline | 17.28 (2.89) | 16.69 (3.82) | 16.88 (3.12)
  Month 12: number analyzed (Participants) | 97 | 84 | 81
  Month 12 | 17.39 (2.73) | 16.46 (3.93) | 16.78 (3.29)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued through the final assessment at Month 12.
Arm/Group | Usual Care | THRIVE App | THRIVE App+Feedback
All-Cause Mortality (participants affected / at risk) | 0/104 | 1/98 | 1/102
Serious Adverse Events (participants affected / at risk) | 15/104 | 9/98 | 6/102
Other Adverse Events (participants affected / at risk) | 2/104 | 0/98 | 1/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=104) | THRIVE App (N=98) | THRIVE App+Feedback (N=102)
Hospitalization (General disorders) | 15 | 9 | 6 — The reason or primary concern for hospitalizations was not collected.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=104) | THRIVE App (N=98) | THRIVE App+Feedback (N=102)
Disease progression caused change in treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Side effects from AET caused change in treatment (Product Issues) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT03592771/Prot_SAP_001.pdf
  • Informed Consent Form (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT03592771/ICF_000.pdf